CLINICAL TRIAL: NCT05456217
Title: Clinical Characteristics and Outcomes of Patients Admitted to Kenyan Critical Care Units During the COVID-19 Pandemic: a Multicenter Registry-based Observational Study
Brief Title: Epidemiological Characteristics and Outcomes of Patients Admitted to Kenyan Critical Care Units (EPOK).
Acronym: EPOK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nat Intensive Care Surveillance - MORU (Other)
Collaborators: Critical Care Society of Kenya (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCAA-K-1-22
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Outcome Studies; Mechanical Ventilation; Kenya

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: admission to ICU — admission to an intensive care unit or high dependency unit in Kenya

SUMMARY:
The Kenyan Critical Care Registry was started in December 2020 and currently involves 10 critical care units in 6 Hospitals. As an initial registry output, we aim to describe patient epidemiological characteristics, initial management and outcomes of critically ill patients in Kenya. This project will provide a much-needed source of clinico-demographic and outcomes data for participating Kenyan critical care units. It will also help to identify processes and outcomes which can be targeted by quality improvement projects, the impact of which can then be evaluated later using the registry.

DETAILED DESCRIPTION:
Background:

The burden of critically ill patients is growing in low and middle income countries (LMICs), but the resources available to assist these patients are limited.1 Critical care is an established and rapidly evolving service in Kenya.2 Yet, patient epidemiological characteristics, patterns of ICU management and patient outcomes in Kenyan ICUs remain scarcely investigated.3,6,7

The ICU registry:

The Kenyan Critical Care Registry was started in December 2020 after receiving ethical approval in November 2020, and currently involves 10 units in 6 Hospitals. The registry was launched in collaboration with the Network for Intensive Care Systems and Training (NICST) and the Mahidol Oxford Research Unit (MORU). As in other countries, the Kenyan Critical Care registry aims to play an increasingly pivotal role in evaluating treatment outcomes, benchmarking services and providing opportunities for service forecasting. Dedicated data collectors in each registry site perform real-time data collection. All registry data is housed and stored securely on a national server located on Kenyan soil. Once entered electronically on password-protected computers at participating facilities, it is automatically encrypted before it leaves the institution for the visualization loop within a ring-fenced server at NICST, where it is unencrypted and aggregated for automated visualization. NICST follows healthcare standard GDP and HIPAA standards. The processed data is then re-encrypted before it is transferred back to the national server, where it is automatically unencrypted and available for review by authorized personnel, through a secure two step log in - a process that is navigated with the help of Kenyan IT teams. An audit trail is created any time the registry is accessed, to see who has logged into it, when, and what data was retrieved or modified.

Study aims:

In this study we aim to describe patient epidemiological characteristics, basic management and outcomes of critically ill patients in Kenya during and after the COVID-19 pandemic, leveraging on the newly-implemented Kenya Critical Care Registry housed under the Critical Care Society of Kenya (CCSK). Study outcomes include clinico-demographic characteristics of patients admitted to critical care units within the Kenya Critical Care Registry network, primary management process measures and short-term critical care outcomes.

Patients:

All patients admitted to participating critical care units from the day of registry onset to the day of database analysis will be included. A secure, non-proprietary, real-time, cloud-based platform designed by NICST, adapted for use at participating facilities when the registry began, is used for data entry and management. A critical care minimum dataset (CCMDS) of variables was employed by the investigators, in consultation with the critical care team at participating facilities.

Ethical Considerations:

Ethical clearance from the Aga Khan University Institutional Ethics Review Committee (IERC) to begin registry creation was obtained in November 2020 (Ref:2019/IERC-89) and a NACOSTI licence secured. Site approvals from NACOSTI-accredited ethical committees and/or administrative clearance were obtained from participating institutions prior to commencement. Ethical/administrative and national regulatory approvals for this present study will be sought in the same manner, prior to study commencement.

Benefits:

There will not be any direct benefit to patients at the outset. The expected improvement in critical care processes and outcomes enabled by the registry data analysis will have the potential to directly benefit future critically ill patients in Kenya. In addition the information gathered on admission, patient flow, occupancy and acuity will be essential to helping Kenyan administrative and management team plan future critical care resource provision, optimising critical care resource utilisation and cost effectiveness. The study may also provide important context specific COVID-19 case-mix and outcome data that may be of value to clinicians, administrators and policy makers during the ongoing pandemic.

Confidentiality:

Access to the electronic registry will be restricted to personnel authorized by the leadership at participating facilities, each of whom have been provided with a unique login and password for this purpose. Each person with such access to the registry has signed a data protection agreement, indicating that they will not share their login details with anyone else, and that they will not share the contents of the registry with unauthorized personnel.

As in other ICU registries, identifiable patient data is restricted to hospital staff authorized to access the critical care registry by the administration of individual facilities.The data extraction for analysis will concern only de-identified data.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an intensive care unit or high dependency unit
* Included in the Kenya Critical Care registry platform

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients admitted to ICUs or HDUs participating in the Kenya Critical Care registry
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 1 month
  death during ICU or HDU stay
Length of ICU stay | 1 month
  duration of stay in the ICU or HDU in days
Demographic characteristics | ICU admission
  The following demographic characteristics are collected: age, sex
APACHE 2 score | ICU admission
  Acute Physiology and Chronic Evaluation 2 score

SECONDARY OUTCOMES:
Patients receiving mechanical ventilation | 1 month
  Proportion of patients receiving invasive mechanical ventilation in the ICU or HDU
Tracheostomy rate | 1 month
  Proportion of patients receiving a tracheostomy in the ICU or HDU
Reason for admission | ICU admission - first 24h
  Reason for admission using APACHE IV classification system and SNOMED CT nomenclature
Use of vasopressors | ICU admission - first 24h
  Use of vasopressors on ICU admission
Use of sedatives | ICU admission - first 24h
  Use of sedative drugs on ICU admission
Use of antibiotics on ICU admission | ICU admission - first 24h
  Proportion of patients with at least one antibiotic prescribed on ICU admission

CONTACTS AND LOCATIONS:
Locations (6):
- Kenya (6):
  - Kisii County Hospital, Kisii
  - Mombasa Aga Khan Hospital, Mombasa
  - Aga Khan University Hospital, Nairobi
  - MP Shah Hospital, Nairobi
  - Nakuru level V Hospital, Nakuru
  - Nyeri County Hospital, Nyeri

REFERENCES:
- [Background] Pisani L, Waweru-Siika W, Sendagire C, Beane A, Haniffa R. Critically ill COVID-19 patients in Africa: it is time for quality registry data. Lancet. 2021 Aug 7;398(10299):485-486. doi: 10.1016/S0140-6736(21)01549-X. No abstract available. PMID 34364515
- [Derived] Njoki C, Simiyu N, Kaddu R, Mwangi W, Sulemanji D, Oduor P, Dona DG, Otieno D, Abonyo TT, Wangeci P, Kabanya T, Mutuku S, Kioko A, Muthoni J, Kamau PM, Beane A, Haniffa R, Dondorp A, Misango D, Pisani L, Waweru-Siika W. EPidemiology, clinical characteristics and Outcomes of 4546 adult admissions to high-dependency and intensive care units in Kenya (EPOK): a multicentre registry-based observational study. Crit Care Explor. 2024 Feb 1;6(2):e1036. doi: 10.1097/CCE.0000000000001036. eCollection 2024 Feb 1. PMID 38356864